CLINICAL TRIAL: NCT02197364
Title: The Role of KL-6 as a Serum Biomarker in the Clinical Diagnosis of Interstitial Lung Diseases (ILD) in China
Brief Title: The Role of KL-6 in the Clinical Diagnosis of ILD
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Principal Investigator, Huiping Li, Professor,Chief of Dept. of Respiratory Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: KL-6_20140715
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Diagnosis; Krebs Von Den Lungen-6
MeSH Terms: conditions — Lung Diseases, Interstitial; Disease; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The residual serums in the clinical laboratory.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ILD, Other respiratory diseases, Healthy control group: ILD: those with interstitial lung disease.
  Other respiratory diseases: those with other respiratory disease including pulmonary tuberculosis, pneumonia, bronchiectasis, chronic obstructive pulmonary disease.
  Healthy control group: those who is healthy.

SUMMARY:
The purpose of the study is to evaluate the significance of KL-6 as a biomarker in the clinical diagnosis of interstitial lung disease (ILD) by detecting serum KL-6 levels among patients with ILD, and comparing them to the clinical diagnostic criteria and other respiratory diseases. In addition, the study discusses the value of KL-6 levels in terms of ILD treatment effect evaluation through the detection of serum KL-6 levels before treatment and after treatment.

DETAILED DESCRIPTION:
As a multi-center, double-blind clinical study, the trial is divided into two parts.

Part 1: The purpose of this part is to evaluate the role of KL-6 as a biomarker in the clinical diagnosis of interstitial lung disease (ILD) by detecting serum KL-6 levels among patients with ILD, and comparing them to the clinical diagnostic criteria and other respiratory diseases, including pulmonary tuberculosis, pneumonia, bronchiectasis, chronic obstructive pulmonary disease and healthy control group.

Part 2: The purpose of this part is to study the value of KL-6 levels in terms of ILD treatment effect evaluation through the detection of serum KL-6 levels before treatment and 30-90 days after treatment. Treatment includes anti fibrosis, anti-inflammatory and other conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Serums from patients with ILD, pulmonary tuberculosis, pneumonia, bronchiectasis, chronic obstructive pulmonary disease and health
* Serums from patients with ILD: before treatment and 30-90 days after treatment

Exclusion Criteria:

* Serums from patients with cancer
* Serums with visible precipitate
* Serums with floc

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The serums from clinical laboratory of Shanghai Pulmonary Hospital, Nanjing Drum Tower Hospital and Beijing Chaoyang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1190 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The KL-6 concentration on the immune analyzer | The serum from patients with ILD will be collected for the duration of hospital stay, an average of 4 weeks
  Detect the KL-6 concentration in serum by the use of the immune analyzer among patients with ILD.

SECONDARY OUTCOMES:
The KL-6 concentration on the immune analyzer | The serum from patients other respiratory diseases will be collected for the duration of hospital stay, an average of 4 weeks
  Detect the KL-6 concentration in serum by the use of the immune analyzer among patients with other respiratory diseases, including pulmonary tuberculosis, pneumonia, bronchiectasis, chronic obstructive pulmonary disease.
The KL-6 concentration on the immune analyzer | The serum from healthy people will be collected for the duration of physical examination, an average of 1 day
  Detect the KL-6 concentration in serum by the use of the immune analyzer among healthy people.
Change of KL-6 concentration on the immune analyzer | pretherapy, 30-90 days after treatment
  Change of KL-6 concentration on the immune analyzer from pretherapy to 30-90 days after treatment among patients with ILD.

CONTACTS AND LOCATIONS:
Overall Officials: Li Hui Ping, Principal Investigator — Shanghai Pulmonary Hospital , Tongji University